CLINICAL TRIAL: NCT03754673
Title: Role of MRI in Diagnosis of Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HMMostafa, Assistant Lecturer, Assiut University
Other Study IDs: Plumonary MRI
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — MRI pulmonary with no contrast administration

SUMMARY:
The aim of this work is to emphasize the role of non-contrast MR imaging in diagnosis of acute pulmonary embolism in comparison to CTA and contrast enhanced MRA as gold standard techniques.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a serious condition responsible for significant morbidity and mortality. PE is currently the third leading cause of cardiovascular death worldwide, so it requires prompt diagnosis and treatment to prevent potentially deadly consequences (1) . Pulmonary embolism occurs when a blood clot-usually from the leg-travels to the lung and blocks the pulmonary artery or one of its branches (2). The diagnosis of acute PE is considered a clinical dilemma due to wide spectrum of multiple nonspecific signs and symptoms (3) .

The D-dimer results are of bad positive laboratory test being positive in other situations rather than PE such as cancer and inflammation (4) .

CT pulmonary angiography (CTA) is highly sensitive and specific for the diagnosis of PE and has become the imaging method of choice in patients suspected of having PE. The multislice CT offered high spatial and temporal resolution imaging in a short time scan. CTA has the ability to assess the pulmonary tree down to the fifth and to eighth order branches in less than 15 seconds due to high speed (5).

However, Limitations of CTPA include exposure to ionizing radiation with its risk of cancer induction and iodinated contrast agent, which carries a risk of allergic reactions and kidney damage and failure in some patients (6) .Many patients with suspected PE, such as pregnant women and patients with impaired renal function, have at least a relative contraindication to contrast media irradiation.

MRI offers a potential alternative to CTPA in the evaluation of the pulmonary vasculature and the diagnosis of PE [7]. To date, however, the majority of studies evaluating the use of MRI in the diagnosis of PE have used gadolinium based intravenous contrast media, which is contraindicated in pregnant patients and in those with renal failure [8].

So, alternatively non contrast MRA improves diagnostic accuracy and simplify the acquisition techniques remains an area of clinically important development. The non-contrast MRA produces enhancing signal from the vessel wall, provides high contrast with no need for bolus timing and provides motion-insensitivity to respiration (9).

The purpose of this study to evaluate the feasibility of detecting pulmonary emboli using non contrast bright blood and dark blood MR imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* High clinical probability of PE assessed by the revised Geneva score and / or had a D- dimer level > 500 µg L1 on an ELISA-based test
* Patients with clinically evident and confirmed by CT PA or contrast enhanced MR-PA to have PE .
* Both sexes will be included in addition to pregnant women.
* No age predilection but children Less than 18 years old will not be included

Exclusion Criteria:

* Patients known to have contraindication for MRI, e.g. an implanted magnetizable device, metallic ocular implant, pacemakers, or claustrophobia.
* Patients with bad general condition with signs of a severe PE such as unstable haemodynamic.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Full history taking and clinical examination.
  2. CT PA or contrast enhanced MR PA.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
detection of pulmonary embolism by MRI without contrast administration | baseline
  diagnosis and detection of pulmonary embolism by MRI in comparison with MSCT pulmonary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Mohammed Mostafa, Asyut, Egypt

REFERENCES:
- [Background] Nyren S, Nordgren Rogberg A, Vargas Paris R, Bengtsson B, Westerlund E, Lindholm P. Detection of pulmonary embolism using repeated MRI acquisitions without respiratory gating: a preliminary study. Acta Radiol. 2017 Mar;58(3):272-278. doi: 10.1177/0284185116651003. Epub 2016 Jul 19. PMID 27273375